CLINICAL TRIAL: NCT01178359
Title: Phase 1 Hospital Based Study of Sodium Nitrite in Resuscitated Cardiac Arrest Patients
Brief Title: Pilot Study of Sodium Nitrite in Resuscitated Cardiac Arrest Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Medic One Foundation (Other)
Responsible Party: Principal Investigator, Francis Kim, Associate Professor, Medicine/Division of Cardiology, University of Washington
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00001499
Record Dates: First submitted 2010-08-06; First posted 2010-08-10 (Estimated); Last update posted 2017-05-18 (Actual); Status verified 2017-05

CONDITIONS: Cardiac Arrest
Keywords: cardiac arrest; ventricular fibrillation; nitrite
MeSH Terms: conditions — Heart Arrest; Ventricular Fibrillation | interventions — Nitrites

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: nitrite

SUMMARY:
Despite advances in cardiac arrest resuscitation survival from cardiac arrest is less than 20-30% and new therapies are urgently needed. Sodium nitrite infused during resuscitation from cardiac arrest has recently been shown to improve survival in a mouse model of cardiac arrest and our group is eager to test this hypothesis in a clinical trial. Our overall hypothesis is that an infusion of 2 μmole/kg sodium nitrite during resuscitation will increase the proportion of patients who will survive cardiac arrest. In preparation for a clinical trial, preliminary safety and efficacy data (phase 1) is needed which is the primary goal of this study.

DETAILED DESCRIPTION:
Sixteen patients will be randomized to receive normal saline (n=5) or doses of IV nitrite (n=11). During the nitrite infusion and for 120 min after the infusion is completed, blood pressure and heart rate will be monitored.

The first 3 patients randomized to receive IV nitrite will receive the lowest dose (1 mg) of IV nitrite and compared to one placebo treated patient. If there is no significant decrease in blood pressure or elevation in heart rate, we will then dose escalate to the 6 mg dose in 4 patients and placebo in two patients. Dose escalation to the highest (14 mg) dose will again be contingent on the absence of significant hypotension or tachycardia in the drug treated patients compared to the pooled (n=3) placebo treated patients. The final block of patients will be randomized to the high nitrite dose (n=4) or placebo (n=2). Final comparisons of all groups will be made to the pooled (n=5) placebo group

ELIGIBILITY:
Inclusion Criteria:

* Successfully resuscitated from cardiac arrest by paramedics in the field Age 18 or older Comatose IV access

Exclusion Criteria:

* traumatic cause of cardiac arrest known DNAR Patient requiring vasopressors at time of randomization SBP <105 PaO2 of less than 90% on FiO2 of 1.0

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2010-01; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Blood pressure | 2 hour
nitrite concentration levels in blood | 2 hour

CONTACTS AND LOCATIONS:
Overall Officials: Francis Kim, MD, Principal Investigator — University of Washington
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States